CLINICAL TRIAL: NCT01834989
Title: Effect of Training and Local Infusion of Insulin-like Growth Factor-I and Training on Tendon Structure in Patients With Patellar Tendinopathy
Brief Title: Patellar Tendinopathy - Effect of Training and Enhancement of the Collagen Synthesis by Insulin-like Growth Factor-I
Acronym: IGF-I
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Principal Investigator, Mette Hansen, Associated Professor, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-4-2012-078
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Tendinopathy
MeSH Terms: conditions — Tendinopathy | interventions — Insulin-Like Growth Factor I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin-like growth factor I (Active Comparator): 3 injection (1 mg), once a week the first 3 weeks of the 12 weeks of intervention
  Interventions: Drug: Insulin-like growth factor I
- Placebo injections (Placebo Comparator): 3 Injections of saline into the patellar tendon 3 times during the first 3 weeks of the 12 weeks interventions period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Insulin-like growth factor I
  Arms: Insulin-like growth factor I
Drug: Placebo
  Other Names: Saline Injections
  Arms: Placebo injections

SUMMARY:
The purpose of the study is to test the hypothesis that stimulation of the synthesis of new structural tendon proteins combined with training improve the tendon structure in patients with chronic knee tendon pain.

DETAILED DESCRIPTION:
Randomized controlled intervention study: 12 weeks intervention period with training and injections of saline or Insulin-Like growth factor I. One year follow-up

ELIGIBILITY:
Inclusion Criteria:

* chronic patellar tendinopathy (> 3 months)
* anterior-posterior thickening of the tendon (1 mm compared to mid-tendon)
* hypo-echoic area with enhanced vascularization

Exclusion Criteria: injection

* corticosteroid injection within the last 12 months
* Knee operation
* Knee osteoarthritis
* Diabetes
* Smoking
* Body mass index >30

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Tendon structure | After 12 weeks intervention (tendon biopsy)

SECONDARY OUTCOMES:
Tendon Pain | 1 year (before and after 12 weeks intervention and 1 year after intervention start)
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjaer, Professor, Principal Investigator — Institute of Sports Medicine, Copenhagen, Bispebjerg Hospital, 2400 Copenhagen, Denmark; Mette Hansen, PhD, Principal Investigator — Section of Sport Science, Department of Public Health, Aarhus University, Dalgas Avenue 4, 8000 Aarhus C, Denmark; Jens Olesen, PhD, Principal Investigator — Institute of Sports Medicine, Copenhagen, Bispebjerg Hospital, 2400 Copenahagen, Denmark
Locations (1):
- Institute of Sports Medicine, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Olesen JL, Hansen M, Turtumoygard IF, Hoffner R, Schjerling P, Christensen J, Mendias CL, Magnusson PS, Kjaer M. No Treatment Benefits of Local Administration of Insulin-like Growth Factor-1 in Addition to Heavy Slow Resistance Training in Tendinopathic Human Patellar Tendons: A Randomized, Double-Blind, Placebo-Controlled Trial With 1-Year Follow-up. Am J Sports Med. 2021 Jul;49(9):2361-2370. doi: 10.1177/03635465211021056. Epub 2021 Jun 17. PMID 34138667
- See also: Study location — http://www.ismc.dk